CLINICAL TRIAL: NCT00259740
Title: An Open-Label, Multi-Center Phase 2 Trial of Denosumab in the Treatment of Relapsed or Plateau-Phase Multiple Myeloma
Brief Title: Open-Label, Phase 2, Proof of Concept Study in Multiple Myeloma - Denosumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050134; NCT00337363 (obsolete NCT alias)
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Results first posted 2011-01-06 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Relapsed or Plateau-Phase Multiple Myeloma
Keywords: Multiple Myeloma, Relapsed, Plateau-Phase
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Denosumab (Experimental)
  Interventions: Drug: DENOSUMAB

INTERVENTIONS:
Drug: DENOSUMAB — 120 mg administered subcutaneously on study days 1, 8, 15, and 29 and every 28 days thereafter. Each dose will be administered in two separate injections of 60 mg (1.0 mL) each.

SUMMARY:
The purpose of this study is to determine if denosumab is effective in the treatment of relapsed or plateau-phase multiple myeloma.

DETAILED DESCRIPTION:
Patients who have relapsed myeloma have failed treatment regimens and have had disease progression following their last treatment regimen. Despite newer salvage therapies, their treatment options are limited and may include best supportive care and investigational therapy. Patients with plateau-phase myeloma have a stabilized serum M-protein level without further tumor regression despite continued treatment. Recent evidence suggests that their prognosis might improve with further reduction in serum M-protein or prolongation of time to disease progression (TTP). These patients are candidates for investigational agents that could further reduce tumor burden or increase TTP.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* clinical diagnosis of relapsed or plateau-phase multiple myeloma
* measurable disease (>0.5 g/dL) as determined by special blood tests
* ECOG 0 or 1

Exclusion Criteria:

* newly diagnosed myeloma
* non-secretory myeloma
* plasma cell leukemia or plasma cell dyscrasia with POEMS syndrome
* prior allogeneic stem cell transplant
* administration of oral or IV bisphosphonates within 2 weeks of enrollment to study

Other criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Vij R, Horvath N, Spencer A, Taylor K, Vadhan-Raj S, Vescio R, Smith J, Qian Y, Yeh H, Jun S. An open-label, phase 2 trial of denosumab in the treatment of relapsed or plateau-phase multiple myeloma. Am J Hematol. 2009 Oct;84(10):650-6. doi: 10.1002/ajh.21509. PMID 19714603
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 13 February 2006 through 8 December 2006
Groups:
- Denosumab 120 mg Q4W - Plateau-Phase: Open-label denosumab 120 mg by subcutaneous injection on day 1 of each 28-day cycle with additional loading doses on days 8 and 15 of cycle 1 in participants with plateau-phase multiple myeloma
- Denosumab 120 mg Q4W - Relapsed: Open-label denosumab 120 mg by subcutaneous injection on day 1 of each 28-day cycle with additional loading doses on days 8 and 15 of cycle 1 in participants with relapsed multiple myeloma
Period: Overall Study
Arm/Group | Denosumab 120 mg Q4W - Plateau-Phase | Denosumab 120 mg Q4W - Relapsed
Started | 43 | 53
Received Study Medication | 42 | 53
Completed | 0 | 0
Not Completed | 43 | 53
Not completed — Physician Decision | 1 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Death | 1 | 1
Not completed — Disease progression | 19 | 36
Not completed — Ongoing | 17 | 3
Not completed — Other | 3 | 0
Not completed — Requirement for alternative therapy | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 120 mg Q4W - Plateau-Phase | Denosumab 120 mg Q4W - Relapsed | Total
Number analyzed (Participants) | 43 | 53 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (11.4) | 62.9 (9.2) | 62.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 13 | 39
  Male | 17 | 40 | 57
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 35 | 39 | 74
  African American | 4 | 7 | 11
  Hispanic or Latino | 1 | 3 | 4
  Other | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Complete Response or Partial Response Based on M-Protein Assessments Only
Description: Complete response or partial response based on serum M-Protein assessments. Complete response is defined as absence of original M-protein in serum by immunofixation, and partial response is defined as ≥ 50% reduction from baseline in serum M-protein, both maintained for a minimum of 6 weeks.
Time Frame: Up to 18 months
Population: All participants who completed the first cycle of treatment with denosumab
Measure: Number; unit: Participants
Arm/Group | Denosumab 120 mg Q4W - Plateau-Phase | Denosumab 120 mg Q4W - Relapsed
Number analyzed (Participants) | 41 | 53
Participants | 0 | 0

2. Secondary Outcome: Complete Response, Partial Response or Minimal Response Based on M-Protein Assessments Only
Description: Complete response, partial response or minimal response based on serum M-protein assessments. Complete and partial responses are as defined for the primary outcome measure. Minimal response is defined as 25 to 49% reduction from baseline in serum M-protein level, maintained for a minimum of 6 weeks.
Time Frame: Up to 18 months
Population: All participants who completed the first cycle of treatment with denosumab
Measure: Number; unit: Participants
Arm/Group | Denosumab 120 mg Q4W - Plateau-Phase | Denosumab 120 mg Q4W - Relapsed
Number analyzed (Participants) | 41 | 53
Participants | 0 | 0

3. Secondary Outcome: Complete Response Based on M-Protein Assessments Only
Description: Complete response based on M-protein assessments, as defined for the primary outcome measure.
Time Frame: Up to 18 months
Population: All participants who completed the first cycle of treatment with denosumab
Measure: Number; unit: Participants
Arm/Group | Denosumab 120 mg Q4W - Plateau-Phase | Denosumab 120 mg Q4W - Relapsed
Number analyzed (Participants) | 41 | 53
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 1 year 6 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Denosumab 120 mg Q4W - Relapsed | Denosumab 120 mg Q4W - Plateau-Phase
Serious Adverse Events (participants affected / at risk) | 14/53 | 6/42
Other Adverse Events (participants affected / at risk) | 38/53 | 32/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg Q4W - Relapsed (N=53) | Denosumab 120 mg Q4W - Plateau-Phase (N=42)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg Q4W - Relapsed (N=53) | Denosumab 120 mg Q4W - Plateau-Phase (N=42)
Anaemia (Blood and lymphatic system disorders) | 8 | 3
Constipation (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 6 | 4
Stomatitis (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 4 | 0
Fatigue (General disorders) | 8 | 8
Oedema peripheral (General disorders) | 0 | 5
Pain (General disorders) | 4 | 0
Pyrexia (General disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4
Sinusitis (Infections and infestations) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 9 | 12
Urinary tract infection (Infections and infestations) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 7
Dizziness (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 4 | 8
Lethargy (Nervous system disorders) | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.